CLINICAL TRIAL: NCT06076551
Title: Sex Difference of Coronary Microvascular Dysfunction Evaluated by Coronary Flow Reserve in Patients With Non-obstructive Coronary Artery Disease
Brief Title: Sex Difference of Coronary Microvascular Dysfunction in Patients With Non-obstructive Coronary Artery Disease
Status: Recruiting | Type: Observational
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Seong-Mi Park, M.D. Ph.D., Professor, Korea University Anam Hospital
Other Study IDs: 2017AN0358
Record Dates: First submitted 2023-09-25; First posted 2023-10-11 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Microvascular Angina
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Adenosine stress echocardiography — Transthoracic echocardiographic assessments will be performed using an ultrasound device (Vivid E95, General Electric Healthcare, Liestal, Switzerland). Color Doppler flow of the distal left anterior descending artery was examined from the modified apical four-chamber view of the anterior interventricular groove. Pulsed-wave Doppler registered blood ﬂow velocity patterns using a sample volume (2-3.0 mm) placed on the color signal. The ultrasound beam was aligned parallel to the vessel ﬂow. The velocity scale of color Doppler was set to 0.21 m/s. Coronary ﬂow Doppler images were acquired at baseline and at 1, 2, and 3 min after adenosine infusion in the same part of the artery. Anti-anginal medications, including calcium channel blockers, were discontinued before the study.

SUMMARY:
Sex difference of coronary microvascular dysfunction evaluated by coronary flow reserve will be assessed in patients with non-obstructive coronary artery disease

DETAILED DESCRIPTION:
The investigators will select consecutive patients who experienced chest pain but had no significant coronary artery stenosis (<50% stenosis). Coronary microvascular function will be evaluated by adenosine stress echocardiography. Coronary blood flow velocities will be measured at 1, 2, and 3 min after adenosine infusion.

Sex difference of coronary microvascular dysfunction evaluated by coronary flow reserve will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Typical/atypical chest pain or ischemic symptoms including dyspnea
* No significant coronary artery stenosis (<50% stenosis) in coronary angiography or computed tomography

Exclusion Criteria:

* ≥ Moderate valvular heart disease
* Congenital heart disease
* Chronic renal failure (estimated glomerular filtration rate <30 ml/min/1.73m2) or end-stage renal failure undergoing hemodialysis or peritoneal dialysis
* Asthma, chronic obstructive pulmonary disease and primary pulmonary hypertension
* Receiving anticancer drugs
* Vasculitis associated with autoimmune diseases
* Atrioventricular block with more than second degrees, symptomatic bradycardia, cryo-node failure syndrome, Wolff-Parkinson-White (WPW) patients

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who experienced chest pain but with no obstructed coronary arteries (<50% stenosis)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite outcome including all-cause mortality, nonfatal myocardial infarction, nonfatal stroke, and hospitalization for heart failure | 1 year
  Number of participants with a composite outcome including all-cause mortality, nonfatal myocardial infarction, nonfatal stroke, and hospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Mi Park, PhD, Principal Investigator — Korea University Anam Hospital; Mi-Na Kim, PhD, Study Chair — Korea University Anam Hospital; Dong-Hyuk Cho, PhD, Study Chair — Korea University Anam Hospital; So Ree Kim, PhD, Study Chair — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No